CLINICAL TRIAL: NCT05040542
Title: A Cohort Study on the Brain Mechanism of Social Emotion and Communication in Infants Aged 0 to 6 Years
Brief Title: The Brain Mechanism of Social Emotion and Communication in Infants Aged 0 to 6 Years
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Xiamen Children's Hospital (Other); ShanghaiTech University (Other); Xi'an Jiaotong University (Other); Shanghai University (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCBN_01
Record Dates: First submitted 2021-07-29; First posted 2021-09-10 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Brain Development; Behavior Disorders, Child; Intellectual Developmental Disorders
Keywords: Preterm; Newborn; Neonates; Infants; Children; Brain; Development
MeSH Terms: conditions — Child Behavior Disorders; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The researchers retain children 2ml serum as a biological sample for the Whole Exon Sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infant Cohort: Healthy infants aged from 0-72 months.This is an observational trial so no intervention will be provided, with exception of study assessments, including fMRI.
  Interventions: Other: maternal exposure during pregnancy

INTERVENTIONS:
Other: maternal exposure during pregnancy — maternal exposure during pregnancy (e.g., environmental exposures and maternal inflammatory states)

SUMMARY:
This study explores the relationship between brain development and infants' social emotion and communication ability, as well as the role of genetic factors and maternal exposure during pregnancy (e.g., environmental exposures and maternal inflammatory states). To provide a theoretical basis for precise intervention of infants' social emotion and communication problems and the overall improvement of brain development.

DETAILED DESCRIPTION:
This study uses functional magnetic resonance imaging (fMRI) is a ultra-fast imaging technology to reflect the changes in brain function when the brain is stimulated or pathologically affected. There are 4 working imaging techniques for fMRI, including blood-oxygen-level dependent fMRI, perfusion weighted imaging (PWI), perfusion weighted imaging (PWI) and MRI spectroscopy. fMRI combine with cloud computing to analyze brain structure, brain function, brain connection, brain development trajectory, multi-modal brain imaging artificial Intelligent calculation, and draw dynamic connection maps of brain development in children aged 0-6 years. In addition, using the Chinese Urban Children's Emotion and Social Assessment Scale (CITSEA) to evaluate children's social and emotional behavior and Gesell Developmental Scale (GDS) to assess the neurological integrity and functional maturity of children, and explore their relationship with brain imaging. The researchers will collect blood samples from the enrollees for whole exome sequencing as well as exposome testing to look for genes related to brain intellectual development and biomarkers related to brain development and to explore their relationship with brain imaging. In addition, the researchers will collect basic information about the family and the mother's health during pregnancy through baseline questionnaires and clinical history data, which will be used to explore pregnancy risk factors for children's brain development and the role of these factors in brain development and the baby's social-emotional and communication skills.

This study explores the relationship between brain development and infants' social emotion and communication ability, as well as the role of genetic factors and maternal exposure during pregnancy (e.g., environmental exposures and maternal inflammatory states). To provide a theoretical basis for precise intervention of infants' social emotion and communication problems and the overall improvement of brain development.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-6 years
2. Born at 34-42 weeks of gestation
3. Birth weight>1500g
4. Normal brain function assessment
5. Parents can understand and sign informed consent

Exclusion Criteria:

1. The mother had severe complications during pregnancy and delivery
2. History of asphyxiation at birth
3. Have congenital structural malformation
4. Have congenital metabolic disease
5. Have major or genetic diseases that affect growth, development or cognition
6. Have contraindications to MRI scanning

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants aged 0-6 years are mainly recruited from the society and Xiamen Children's Hospital.
Sampling Method: Probability Sample
Enrollment: 3001 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Brain structure (cortical thickness) change of subjects | at baseline,and 6 months after baseline.
  Using T1 weighted and T2 weighted images to measure brain cortical thickness, analyzing the brain structural changes (differences of cortical thickness) over time.
Brain structural connectivity change of subjects | at baseline,and 6 months after baseline.
  Using diffusion-weighted images to measure the structural connectivity matrix (based on fiber tracking) of brain, analyzing the brain structural connectivity changes (differences in fibers number) over time.
Brain functional connectivity change of subjects | at baseline,and 6 months after baseline.
  Using resting state functional MRI (blood-oxygen-level dependent) to measure the functional connectivity matrix, analyzing the brain functional connectivity (differences in connectivity strength) changes over time.
Cerebral blood flow change of subjects | at baseline,and 6 months after baseline.
  Using arterial spin labeling (ASL) to measure relative cerebral blood flow (rCBF) can produce quantitative cerebral perfusion images, analyzing the change (differences in rCBF) of brain perfusion over time.
EEG examination change of subjects | at baseline, and 6 months after baseline.
  EEG data were collected at each follow-up visit. Electroencephalogram (EEG), especially the event-related potential (ERP) technique, can non-invasively explore the cognitive processes of infant speech recognition, language comprehension, phonological awareness, recognition memory, and facial emotion recognition. The study will collect EEG data from children in resting states, including the power spectral density of different frequency bands (e.g., delta, theta, alpha, beta, gamma), ERP waveform, amplitude, and latency during specific cognitive or sensory tasks, and EEG network connectivity in resting and task states. Through an experimental paradigm designed specifically for different age groups, the influential factors of language and social-emotional development in 0-3 years old infants were explored.
Social and emotional behavior change of subjects (CITSEA score) | at baseline,and 6 months after baseline.
  Using Chinese Version of Urban Infant-Toddler Social and Emotional Assessment (CITSEA) to evaluate children's social and emotional behavior, including four broad domains: 1) externalizing problems; 2) internalizing problems; 3) dysregulation problems; 4) competencies. The problem behavior domain T score >63 is assessed as suspicious positive, indicating possible social-emotional behavior problems; the competencies domain T score <37 is assessed as suspicious positive, indicating there may be a delay in the development of social-emotional ability, analyzing the CITSEA score changes over time.
Brain development change of subjects (GDS score) | at baseline,and 6 months after baseline.
  Using Gesell Development Scale (GDS) to assess neurological integrity and functional maturity of children, including adaptive behavior, gross motor behavior, fine motor behavior, language behavior and personal social behavior. Mild intellectual disability: 55≤DQ≤75; moderate intellectual disability: 40≤DQ≤54; severe mental disability:25≤DQ≤39; extreme intellectual disability: DQ<25, analyzing the GDS score changes over time.
Developmental level prediction change of subjects (brain age, CITSEA and GDS score) | at baseline,and 6 months after baseline.
  Using a connectome-based predictive model (CPM) to predict the developmental levels of subjects. In the modal training procedure, extracted multimodal MRI measures (primary outcomes 1 to 4) are input features, and the age, CITSEA and GDS score are ground truths.
Child behavioral development change of subjects | at baseline,and 6 months after baseline.
  Griffiths Development Scales - Chinese Edition (GDSC) : Griffith scale in Chinese children aged 0 ~ 8 speakers of standardized rating scale, with Chinese standard. The scale is divided into two parts, 0-2 years old and 0-8 years old. The 0-2 years old part is composed of 5 fields: The 0-2 years old part is composed of 5 fields, such as "A action ", "B individual-social ", "C language ", "D hand-eye coordination "and "E performance", and the 0-8 years old part adds "F practical reasoning field "on this basis. When the development quotient DQ<70, development is delayed, and when DQ≥85, development is normal.
Child mental health change of subjects | at baseline, and 6 months after baseline.
  Ages and Stages Questionnaires: Social-Emotional, Second Edition (ASQ:SE-2) : This scale is used to assess a child's social-emotional development. In general, a higher score means a child needs more attention or is in a higher risk state for social-emotional development.
Intelligence quotient change of subjects | at 3 years old, 4 years old, 5 years old, and 6 years old.
  Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV) : Use the Chinese version (revised by Professor Zhang Houcan) to assess children's intelligence level. Choose 10 core tests and 4 auxiliary tests from WISC-IV. Four scores, namely the Verbal Comprehension index (VCI), Perceptual Reasoning Index (PRI), Working memory Index (WMI), and processing speed Index (PSI), were calculated from the question bank, and the four composite scores were recombined to form the General Ability Index (GAI) and Cognitive Ability Index (CPI). The resulting total Intelligence quotient (FSIQ). A FSIQ score between 85 and 115 is considered normal intelligence; Between 70 and 84 are classified as borderline intelligence; Less than 70 is classified as low intelligence.

SECONDARY OUTCOMES:
Biomarker Screening | one time blood draw at baseline.
  At enrollment, 0.5 ml of blood was drawn from each parent and child for the exposome. High - throughput sequencing technology will be used to screen for biomarkers associated with brain development.
Relationship Assessment between Biomarkers and Development | at baseline.
  The relationship between the identified biomarkers and children's cognitive and emotional development will be assessed. This will provide a database for understanding the relationship between environment and development, and a scientific basis for future intervention strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Deyi Zhuang, Dean, Study Chair — Xiamen Children's Hospital
Locations (1):
- Xiamen Children's Hospital, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ball G, Pazderova L, Chew A, Tusor N, Merchant N, Arichi T, Allsop JM, Cowan FM, Edwards AD, Counsell SJ. Thalamocortical Connectivity Predicts Cognition in Children Born Preterm. Cereb Cortex. 2015 Nov;25(11):4310-8. doi: 10.1093/cercor/bhu331. Epub 2015 Jan 16. PMID 25596587
- [Background] Cao M, He Y, Dai Z, Liao X, Jeon T, Ouyang M, Chalak L, Bi Y, Rollins N, Dong Q, Huang H. Early Development of Functional Network Segregation Revealed by Connectomic Analysis of the Preterm Human Brain. Cereb Cortex. 2017 Mar 1;27(3):1949-1963. doi: 10.1093/cercor/bhw038. PMID 26941380
- [Background] Cao M, Huang H, He Y. Developmental Connectomics from Infancy through Early Childhood. Trends Neurosci. 2017 Aug;40(8):494-506. doi: 10.1016/j.tins.2017.06.003. Epub 2017 Jul 3. PMID 28684174
- [Background] Emerson RW, Adams C, Nishino T, Hazlett HC, Wolff JJ, Zwaigenbaum L, Constantino JN, Shen MD, Swanson MR, Elison JT, Kandala S, Estes AM, Botteron KN, Collins L, Dager SR, Evans AC, Gerig G, Gu H, McKinstry RC, Paterson S, Schultz RT, Styner M; IBIS Network; Schlaggar BL, Pruett JR Jr, Piven J. Functional neuroimaging of high-risk 6-month-old infants predicts a diagnosis of autism at 24 months of age. Sci Transl Med. 2017 Jun 7;9(393):eaag2882. doi: 10.1126/scitranslmed.aag2882. PMID 28592562
- [Background] Emerson RW, Gao W, Lin W. Longitudinal Study of the Emerging Functional Connectivity Asymmetry of Primary Language Regions during Infancy. J Neurosci. 2016 Oct 19;36(42):10883-10892. doi: 10.1523/JNEUROSCI.3980-15.2016. PMID 27798142
- [Background] Tavor I, Parker Jones O, Mars RB, Smith SM, Behrens TE, Jbabdi S. Task-free MRI predicts individual differences in brain activity during task performance. Science. 2016 Apr 8;352(6282):216-20. doi: 10.1126/science.aad8127. Epub 2016 Apr 7. PMID 27124457
- [Background] Zhang Y, Shi F, Wu G, Wang L, Yap PT, Shen D. Consistent Spatial-Temporal Longitudinal Atlas Construction for Developing Infant Brains. IEEE Trans Med Imaging. 2016 Dec;35(12):2568-2577. doi: 10.1109/TMI.2016.2587628. Epub 2016 Jul 7. PMID 27392345
- [Background] Zhang W, Li R, Deng H, Wang L, Lin W, Ji S, Shen D. Deep convolutional neural networks for multi-modality isointense infant brain image segmentation. Neuroimage. 2015 Mar;108:214-24. doi: 10.1016/j.neuroimage.2014.12.061. Epub 2015 Jan 3. PMID 25562829
- [Derived] Huang X, Su C, Lin Y, Zhou T, Ye R, Li D, Liu M, Wu G, Li W, Xie N, Deng X, Zhu N, Lin S, Li Q, Yan K, Zhuang D. Cohort protocol: risk assessment of maternal inflammation and early brain development in infants and young children based on multi-source data modeling. Front Public Health. 2025 Jul 14;13:1530285. doi: 10.3389/fpubh.2025.1530285. eCollection 2025. PMID 40726941
- [Derived] Xu X, Wang Z, Zhang W, Guo J, Wei W, Zhang M, Ding X, Liu X, Yang Q, Wang K, Zhu Y, Sun J, Song H, Shen Z, Chen L, Shi F, Wang Q, Li Y, Zhang H, Li D. Behavioral observation and assessment protocol for language and social-emotional development study in children aged 0-6: the Chinese baby connectome project. BMC Psychol. 2024 Oct 4;12(1):533. doi: 10.1186/s40359-024-02031-x. PMID 39367488